CLINICAL TRIAL: NCT03474133
Title: Brentuximab Vedotin as Alternative to the Autologous Stem Cell Transplantation in Relapsed and Refractory Classical Hodgkin's Lymphoma (BASALT)
Acronym: BASALT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Basalt001
Record Dates: First submitted 2018-03-12; First posted 2018-03-22 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's lymphoma; Hodgkin lymphoma; relapsed; refractory; brentuximab vedotin; autologous stem cell transplantation
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brentuximab (Experimental): Brentuximab vedotin 1,8 mg/kg, every 21 days, up to 16 cycles
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — brentuximab vedotin 1,8 mg/kg, intravenous infusion every 21 days, up to 16 infusions per patient during study period
  Other Names: Adcetris

SUMMARY:
This study evaluate possibility of brentuximab vedotin, administered after first treatment failure (no response or relapse after I line therapy) of Hodgkin's lymphoma, to induce durable response or cure without autologous stem cell transplantation.

DETAILED DESCRIPTION:
Brentuximab vedotin (BV) can induce durable response or cure in some patients with relapsed or refractory Hodgkin's lymphoma (RR HL) after autologous stem cell transplantation (ASCT) failure. It is expecting that BV alone administered earlier (after first treatment failure, without any additional treatment) can cure some RR HL patients and spare them from ASCT-associated risks and toxicity. Therefore in this study full course of BV which confirmed its curative potential in post-ASCT setting will be applicated to the potentially transplant-eligible RR HL patients immediately after first treatment failure, with a aim to assess curative potential of BV in this setting.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years or older
2. Voluntary written informed consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
3. Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
4. Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
5. Patients must have a diagnosis of a morphologically confirmed cluster of differentiation antigen 30 {CD30)-positive classical Hodgkin's lymphoma with primary refractory course or relapse after adequate first-line chemotherapy (with morphologically confirmation of vital tumor)
6. PET-positive measurable disease (at least one lesion with Deauville score of >3 and at >1.5 cm on CT scan)
7. Performance status Eastern Cooperative Oncology Group (ECOG) <3
8. Patients potentially eligible for subsequent ASCT according treating physician decision
9. Clinical laboratory values as specified below within 7 days before the first dose of study drug:

   * Absolute neutrophil count ≥ 1,500/µL unless there is known hematologic/solid tumor marrow involvement
   * Platelet count ≥ 75,000/ µL unless there is known marrow involvement of the disease
   * Total bilirubin must be < 1.5 x the upper limit of the normal (ULN) unless the elevation is known to be due to Gilbert syndrome.
   * ALT or aspartate aminotransferase (AST) must be < 3 x the upper limit of the normal range. AST and ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of HL tumor in liver.
   * Serum creatinine must be < 2.0 mg/dL and/or creatinine clearance or calculated creatinine clearance > 40 mL/minute.
   * Hemoglobin must be ≥ 8g/dL.

Exclusion Criteria:

1. More than one line of chemotherapy due to Classical Hodgkin's lymphoma (any salvage treatment)
2. Previous treatment with brentuximab vedotin
3. Female patient who are both lactating and breast-feeding or have a positive serum pregnancy test during the screening period
4. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol.
5. Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of progressive multifocal leukoencephalopathy (PML)
6. Symptomatic neurologic disease compromising normal activities of daily living or requiring medications
7. Any sensory or motor peripheral neuropathy greater than or equal to Grade 2
8. Known history of any of the following cardiovascular conditions

   * Myocardial infarction within 2 years of enrollment
   * New York Heart Association (NYHA) Class III or IV heart failure (see appendix #1)
   * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
   * Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50%
9. Any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first study drug dose
10. Patients that have received other investigational agents within at least 5 half-lives of last dose of that prior treatment
11. Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin.
12. Known human immunodeficiency virus (HIV) positive
13. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
14. Diagnosed or treated for another malignancy. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Continuous complete response (CCR) rate | 3 years
  Rate of complete responses lasting without further treatment at least 3 years after initiation of BV therapy

SECONDARY OUTCOMES:
Additional therapy-free survival (ATFS) | 3 years
  time from the first dose of study medication to one of the following events: unsatisfactory investigational treatment effect (as defined as Deauville score >3 on first positron emission computed tomography/ computer tomography (PET/CT) and >2 on second), progression or relapse, death of any cause or initiation of any additional anti-lymphoma therapy (except consolidation radiotherapy) without confirmed unsatisfactory investigational treatment effect, progression or relapse
Overall survival | 3 year
  time from the first dose of BV to the death of any cause
Incidence AE according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 [Safety] | 1 year
  incidence AE according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay Zhukov, MD, Phd, Principal Investigator — Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology
Locations (2):
- Russia (2):
  - City clinical hospital №40, Moscow
  - R. Gorbacheva Research Institute of Pediatric Hematology and Transfusiology; Pavlov State Medical University of Saint-Petersburg, Saint Petersburg